CLINICAL TRIAL: NCT05426694
Title: Effectiveness of Scapular Clock Exercises in Scapular Dyskinesia; A Randomized Clinical Trial
Brief Title: Effectiveness of Scapular Clock Exercises in Scapular Dyskinesia in Post-Operative Open Heart Surgery Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Faisalabad (Other)
Responsible Party: Principal Investigator, Sana Zahir, Dr Sana Zahir;PT and Dr Aqsa Shahid;PT, University of Faisalabad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TUF/DR/DPT/366
Record Dates: First submitted 2022-05-25; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Scapular Dyskinesis
Keywords: Scapular dyskinesia; Scapular Clock Exercises; Open Heart Surgery
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: There were 30 subjects divided equally and randomly into Group A and Group B. Group A was receive the intervention while group B will be active control group. The duration of treatment will be equal for both groups, that is 3 sessions per week for a period of 4 weeks.
Who Masked: Participant
Masking Description: Only the participants were masked. They did not know either they are in the interventional group or in the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): The interventional group received stretching and strengthening exercises along with scapular clock exercises. For the first two weeks, only scapular clock exercises were performed by the patient actively. After 2 weeks, the subjects performed scapular clock exercises by using the thera-band.
  Interventions: Other: Scapular clock exercises; Other: Stretching and strengthening exercises
- Group B (Active Comparator): The active control group received stretching and strengthening exercises only. The stretching and strengthening exercises include corner stretch, wall-washes and pectoralis minor muscle stretch.
  Interventions: Other: Stretching and strengthening exercises

INTERVENTIONS:
Other: Scapular clock exercises — In scapular clock exercises, the hand is placed on the wall in front of your body. Move the hand in direction of 12 and 6 o'clock to elevate and depress the scapula. Then move hands towards 9 o' clock and 3 o'clock direction to protract and retract the scapula. Hold each position for 10 seconds. From 3rd week and onward the patient will use thera-band and then perform clock exercises.
  Other Names: Stretching and strengthening exercises (Physical Therapy)
  Arms: Group A
Other: Stretching and strengthening exercises — Stretching and strengthening exercises of shoulder and scapular muscles was performed including wall washes, corner stretch, pectoral muscles stretch and wall push ups.

SUMMARY:
In patients after open-heart surgery, the complaint of scapular dyskinesia is very common. It occurs due to the weakness of the muscles surrounding the scapula. In this research, investigators checked the effectiveness of scapular clock exercises in scapular dyskinesia, in post-op open heart surgery patients. There were two groups, an intervention "Active group" and a 'control group'. The patients will be randomly assigned to each group equally. The treatment session was given for a period of 4 weeks, with 3 sessions each week. They were assessed before treatment, after 2 weeks and post-intervention.

DETAILED DESCRIPTION:
Scapular dyskinesia is the malalignment of the scapula. It occurs when the pectoralis muscle (pectoralis minor) becomes tight and there is the weakness of the trapezius muscle (lower fibers). It can commonly occur after open-heart surgery due to incision and prolonged bed rest. In this research, the effectiveness of scapular clock exercises was checked. These exercises can strengthen the weak trapezius muscle and also stretch the tight pectoralis minor muscle. By adding these exercises in cardiac rehabilitation the occurrence of scapular dyskinesia can be reduced. Post-op open heart surgery patients mostly present with complain of shoulder pain. Most of their treatment is directed towards shoulder joint while the scapula is usually ignored. So it is important to add exercises directed towards the scapula along with shoulder.

In this study, The investigators will recruit 30 post-op cardiac surgery patients with complain of shoulder pain, with positive scapular dyskinesia. The sample size was calculated using formula and the values were taken from previous researches. Scapular assistance test and Scapular retraction test was used to find out patients with scapular dyskinesia. The subjects will then be randomly divided into two groups using online randomization generator. The interventional group was receive stretching and strengthening exercises with additional scapular clock exercises and the active control group will receive stretching and strengthening exercises. There was 3 sessions per week, for a period of 4 weeks. The patients was assessed prior to the treatment , then after 2 weeks and later after completion of 4 weeks. The tools for assessment include NPRS for pain, Quick-DASH for activity limitation of shoulder and goniometer for measuring range of motion of shoulder.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose open heart surgery is done at least 6weeks ago.
* Subjects having shoulder and scapular region pain.
* 50% or less loss of Active ROM of shoulder in abduction, flexion and external rotation.
* Positive Scapular assistance (SAT) and Scapular retraction test.
* Positive findings on observational examination of scapula, showing abnormal prominence of either inferior, medial or superior border of scapula.
* Type I and Type II scapular dyskinesia present
* Consented to take part in the study.

Exclusion Criteria:

* • Bilateral shoulder involvement

  * History of previous surgery on shoulder
  * Shoulder fracture
  * Glenohumeral or acromioclavicular joint Arthritis.
  * Neuromuscular disorders

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-06-20 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Shoulder pain | 4 weeks
  Shoulder pain was assessed by using the Numeric Pain Rating (NPRS) Scale. NPRS is an 11-item Likert scale having 0 as no pain and 10 as maximum pain

SECONDARY OUTCOMES:
Level of Shoulder activity limitation | 4 weeks
  The level of shoulder activity limitation was assessed by using the Quick-DASH questionnaire. There were 11 questions that were rated by the Likert scale having 1 as no disability and 5 as maximum disability

OTHER OUTCOMES:
Shoulder Range of Motion (ROM) | 4 weeks
  Shoulder ROM will be assessed by using a Goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Izza Ayub, MS Physical Therapy, Principal Investigator — The University of Faisalabad
Locations (1):
- Faisalabad Institute of Cardiology, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No